CLINICAL TRIAL: NCT00844077
Title: Preliminary Longitudinal Validation of Biomarkers Predictive of Barrett's Esophagus Progression to Dysplasia and Adenocarcinoma
Brief Title: Preliminary Longitudinal Validation of Biomarkers Predictive of Barrett's Esophagus
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Early Detection Research Network (Network); M.D. Anderson Cancer Center (Other); Unity Health Toronto (Other); Dana-Farber Cancer Institute (Other); Dartmouth-Hitchcock Medical Center (Other); Columbia University (Other); Icahn School of Medicine at Mount Sinai (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Missy Tuck, Project manager, Clinical Trials, University of Michigan
Other Study IDs: GLNE 008; 5U01CA086400-08 (NIH)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Intestinal Metaplasia
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma,serum, DNA, urine, Barrett's tissue (Fixed and Frozen), Normal Esophagus tissue (Fixed and Frozen)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Barrett's metaplasia: Barrett's intestinal metaplasia, confirmed via pathology, undergoing standard of care endoscopic screening.

SUMMARY:
Barrett's esophagus can progress to esophageal cancer, but it doesn't always. Current treatment is frequent surveillance via upper endoscopy with multiple biopsies to look for changes (dysplasia). Pathologists vary dramatically in their interpretation of Barrett's Metaplasia versus dysplasia and consensus is very difficult to achieve. The investigators propose a longitudinal study of subjects with confirmed Barrett's intestinal metaplasia without dysplasia to look for predictive factors for transformation to dysplasia or cancer. Potential biomarkers can be found in serum, plasma, urine, frozen or fixed Barrett's and Normal esophageal mucosa. In addition, the investigators are testing a brushing technique from CDx, Inc. for predictive factors. Subjects must have pathologically confirmed Barrett's intestinal metaplasia without history of dysplasia to be on this longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old)
* Subjects with pathologically confirmed Barrett's esophagus, including:
* Intestinal metaplasia without dysplasia, long and short segments (>1 cm)
* Intestinal metaplasia without dysplasia, long and short segments (>1 cm), previously in GLNE 003
* Intestinal metaplasia without dysplasia with indefinite-for-dysplasia (or history of indefinite-for-dysplasia) provided there is no history of HGD, or EAC.
* Intestinal metaplasia without dysplasia or indefinite-for-dysplasia with a history of LGD provided the last surveillance endoscopy showed IM alone, the LGD history was at least 12 or more months ago and there is no history of HGD or EAC.
* Able to physically tolerate removal of 34 ml of blood
* Tolerate extra research related biopsies and brushings
* Willing to permit extra biopsies at future endoscopic procedures
* Ability and willingness to complete questionnaires
* Willing to sign informed consent Exclusion Criteria
* Subjects with a pathologically confirmed history of Barrett's, HGD or EAC
* Subjects with pathologically confirmed history of Barrett's LGD within the last 12 months.
* Subjects in whom esophageal biopsy would be contraindicated (eq. varices)
* Subjects with serious infections requiring IV antibiotics
* Subjects with known HIV or chronic viral hepatitis
* Subjects on active chemotherapy or radiation treatment
* Subjects who have had an esophagectomy
* Subjects with an active malignancy diagnosed or treated within 3 years except for squamous cell carcinoma of the skin, basal cell carcinoma of the skin; Carcinoma in situ, Stages Ia or Ib invasive squamous cell carcinoma of the cervix treated by surgery and/or radiation therapy; Stage Ia Grade 1 adenocarcinoma of the endometrium treated with surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing clinically-indicated upper endoscopy for surveillance of their pathologically-confirmed Barrett's intestinal metaplasia. Recruitment is from the Endoscopy schedules of the collaborating locations.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2007-10; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Conversion from Barrett's intestinal metaplasia to dysplasia or esophageal adenocarcinoma. | 5-8 years

CONTACTS AND LOCATIONS:
Overall Officials: Dean E Brenner, MD, Principal Investigator — University of Michigan
Locations (6):
- United States (5):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- St. Michael's Hospital, Toronto, Ontario, Canada